CLINICAL TRIAL: NCT04239287
Title: Lung Function and Exercise Response Measured by Optoelectronic Plethysmography in School-aged Children Born Preterm
Brief Title: Preterm Lung Function and Exercise Response Measured by OEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Northumbria University (Other)
Responsible Party: Sponsor
Other Study IDs: 09040
Record Dates: First submitted 2019-10-01; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Premature Birth
Keywords: Lung function; Exercise
MeSH Terms: conditions — Premature Birth; Motor Activity | interventions — Respiration; Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm: Children age 8-16 years born at <32 weeks gestation.
  Interventions: Diagnostic Test: Lung function + exercise tests
- Control: Children age 8-16 years born at >37 weeks gestation
  Interventions: Diagnostic Test: Lung function + exercise tests

INTERVENTIONS:
Diagnostic Test: Lung function + exercise tests — Lung function + exercise tests

SUMMARY:
This study will explore lung function and respiratory health in school-aged children who were born prematurely at <32 weeks gestation. It will involve full lung function assessment, a questionnaire and discussion about respiratory health, and an exercise test using optoelectronic plethysmography (OEP) to measure breathing patterns.

DETAILED DESCRIPTION:
Preterm are born during a critical stage of lung development, and can have abnormalities in lung function that persist with age. Previous studies have shown that children with BPD have reduced lung function and limited exercise capacity. These studies have used conventional lung function testing which requires a tight fitting mask. This is uncomfortable, may alter normal breathing patterns and cannot measure changes in total lung volume.

Optoelectronic plethysmography (OEP) indirectly measures lung volumes and breathing patterns using cameras to track the position of marker stickers on the chest, back and abdomen. It is comfortable, does not require a mask and allows us to track changes in total lung volume.

This study will use standard lung function testing and OEP to measure lung function and breathing patterns at rest and during exercise in school-aged children born prematurely, compared to healthy children born at full term. All participants will complete standard lung function tests, a questionnaire and structured interview to qualitatively assess respiratory health, and an exercise test using OEP to assess how breathing changes with exercise.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-16 years
* Born at <32 weeks gestation (preterm) or >37 weeks gestation (controls)
* Parental consent obtained

Exclusion Criteria:

* Unable to comply with test procedure
* Respiratory illness within last 2 weeks
* Cardiac disease (excludes ligated PDA)
* Neuromuscular disease

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm participants will be aged 8-16 years, and previously admitted to the neonatal unit at the Royal Victoria Infirmary, Newcastle upon Tyne.
  Controls will be healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-09-02 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in end-expiratory lung volume with exercise | Pre + post exercise (10minutes)
  Change in end-expiratory lung volume measured in litres with exercise measured using optoelectronic plethysmography

SECONDARY OUTCOMES:
Change in tidal volume with exercise | During exercise (10 minutes)
  Change in tidal volume with exercise measured in litres using optoelectronic plethysmography
Change in minute ventilation with exercise | During exercise (10 minutes)
  Change in minute ventilation (measured in litres/minute) with exercise measured using optoelectronic plethysmography.
Baseline forced expiratory volume in 1 second (FEV1) | Baseline
  Baseline forced expiratory volume (in litres) in 1 second measured by spirometry (FEV1)
Forced vital capacity (FVC) | Baseline
  Baseline forced vital capacity measured in litres (FVC)
Forced mid-expiratory flow (FEF25-75%) | Baseline
  Mean forced expiratory flow between 25% and 75% of FVC measured in litres/second (FEF25-75%)
Transfer factor for carbon monoxide (TLCO) | Baseline
  Transfer factor for carbon monoxide (measured in millimoles per minute per kilopascal) using single breath test
Body plethysmography | Baseline
  Baseline lung volume (in litres) measured using body plethysmography
FeNO | Baseline
  Baseline FeNO (fraction of exhaled nitric oxide)
Exercise induced bronchoconstriction | 10 minutes post exercise
  % change in FEV1
Baseline activity levels | 1 week period
  Baseline activity levels measured using Actigraph monitor

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J O'Brien, MBBS, Principal Investigator — Newcastle upon Tyne Hospitals NHS Foundation Trust
Locations (1):
- Royal Victoria Infirmary, Newcastle, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided